CLINICAL TRIAL: NCT00885066
Title: Phase I Study of Gemcitabine, Capecitabine, and Erlotinib Together in Advanced Pancreatic Cancers
Brief Title: Gemcitabine, Capecitabine, and Erlotinib in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/36; CALACASS-CAPERGEM; ROCHE-CALACASS-CAPERGEM; INCA-RECF0622; 2007-005072-14 (EudraCT Number)
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2015-02

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Erlotinib Hydrochloride; Gemcitabine

ARMS (1):
- gemcitabine, capecitabine, erlotinib (Experimental)
  Interventions: Drug: capecitabine; Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine
Drug: erlotinib hydrochloride
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of gemcitabine given together with capecitabine and erlotinib in treating patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum-tolerated dose of the combination of gemcitabine hydrochloride, capecitabine, and erlotinib hydrochloride in patients with advanced pancreatic cancer.

Secondary

* Analyze the limiting toxicities according to CTC.
* Analyze the toxicity according to CTC.
* Determine the recommended dose.
* Determine the pharmacokinetic dosages of the three drugs.
* Analyze interactions between the drugs.

OUTLINE: This is a multicenter study.

Patients receive one course of chemotherapy comprising gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, oral capecitabine twice daily on days 1-21, and oral erlotinib hydrochloride once daily on days 1-28.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Advanced disease
* No standard curative therapy available
* Must have received prior first-line chemotherapy
* No brain metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 8 weeks
* ANC ≥ 1.5 x 10^9/ L
* Platelet count ≥ 130 x 10^9/ L
* Hemoglobin ≥ 10 g/dL
* Liver transaminases ≤ 1.5 times upper limit of normal (ULN) (≤ 5 times ULN in the presence of liver metastases)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 130 mmol/L OR creatinine clearance > 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No intolerance or hypersensitivity to any of the drugs being tested
* No history of interstitial lung disease
* No history of severe cardiac disease
* No serious uncontrolled infection
* No rare hereditary disorders, i.e., galactosemia, lactase deficiency, or malabsorption of glucose or galactose syndrome
* Must not be deprived of liberty or under guardianship
* Must not be on probation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior erlotinib hydrochloride
* No concurrent potent inducers or inhibitors of cytochrome P450 or CYP3A4
* More than 14 days since participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Clinical or laboratory toxicities as assessed by CTC | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Francois, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France